CLINICAL TRIAL: NCT01751204
Title: A Randomized, Double-blind, Crossover Study to Compare the Absorbability Between Calcium Tablet and Calcium Ion Water
Brief Title: Comparison of Absorbability Between Calcium Tablet and Calcium Ion Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: CHUGOKU KAYAKU CO., LTD. (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-677
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcium tablet (Active Comparator): 250 mg calcium/tablet
  Interventions: Dietary Supplement: Calcium tablet
- Calcium ion water (250mg) (Experimental): 250 mg calcium in 200 ml water
  Interventions: Dietary Supplement: Calcium ion water (250mg)
- Calcium ion water (125mg) (Experimental): 125 mg calcium in 200 ml water
  Interventions: Dietary Supplement: Calcium ion water (125mg)

INTERVENTIONS:
Dietary Supplement: Calcium tablet
  Arms: Calcium tablet
Dietary Supplement: Calcium ion water (250mg)
  Arms: Calcium ion water (250mg)
Dietary Supplement: Calcium ion water (125mg)
  Arms: Calcium ion water (125mg)

SUMMARY:
The purpose of this study is to evaluate the absorbability of calcium tablet and calcium ion water.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females

Exclusion Criteria:

* Taking medicines or functional food that affect serum calcium levels
* Diseases that affect bone
* Renal or hepatic dysfunction
* Heart disease
* Participation in any clinical trial within 90 days of the commencement of the trial

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Serum calcium profile (including AUC, Cmax, and Tmax) | Overall 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan